CLINICAL TRIAL: NCT01073332
Title: Arginine and Antioxidant Supplement on Performance in Elderly Male Cyclists: A Randomized Controlled Trial
Brief Title: The Effects of a Dietary Supplement on Exercise Performance in Healthy Older Adults"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UCLA_IRB_03-08-087-01
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2010-02

CONDITIONS: Excessive Physical Exercise, Unspecified

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo group received a powder with all active ingredients replaced with M-100 maltodextrin.
  Interventions: Dietary Supplement: Placebo
- Arginine antioxidant supplements (Experimental): Dietary Supplement: Niteworks
  Interventions: Dietary Supplement: Arginine antioxidant supplements

INTERVENTIONS:
Dietary Supplement: Arginine antioxidant supplements — The proprietary supplement Niteworks® was manufactured by Herbalife International Inc. (Century City, California, USA). Each serving contained 5.2g L-arginine in a proprietary blend with L-citrulline, 500mg ascorbic acid, 400IU vitamin E, 400ug folic acid, 300mg L-taurine, and 10mg alpha lipoic acid in a lemon-flavored powder form. One serving of supplement powder was mixed with 8 oz of water, administered at bedtime based on the rationale that nitric oxide levels are lowest during sleep due to inactivity, lack of food and low blood pressure.
  Arms: Arginine antioxidant supplements
Dietary Supplement: Placebo — The placebo group received a powder with all active ingredients replaced with M-100 maltodextrin.
  Arms: Placebo

SUMMARY:
Human exercise capacity decreases with aging. One explanation may be that blood vessels stiffen with age and release less of a compound called nitric oxide (NO). This compound normally relaxes blood vessels and increases blood flow to muscles, but damaging compounds called free radicals can interfere with this process. Antioxidants may help prevent free radicals from inactivating nitric oxide. The purpose of this study was to investigate the effects of an antioxidant supplement that supports NO production on exercise performance in elderly male cyclists.

DETAILED DESCRIPTION:
Since the discovery of the vascular smooth muscle relaxant properties of nitric oxide (NO) over 25 years ago, studies have implicated this molecule in modulating such processes as atherosclerosis, impotence, angina, platelet function, and blood pressure, among others. Through vascular smooth muscle relaxation in both coronary and skeletal muscle arteries, as well as via independent mechanisms, nitric oxide has also been implicated in improvement of exercise capacity. In addition, NO may be involved in the immune system, assist in memory function and sleep regulation, and act as a cellular signaling messenger. Youthful, healthy and athletic individuals generally have a healthier NO system, compared to sedentary, unhealthy and aging individuals. NiteworksTM is a dietary supplement that includes L-arginine, an amino acid that acts as a nitric oxide donor and has been shown to increase levels of this molecule in the body. NiteworksTM has been formulated as a composite mixture along with other supplements, including antioxidants, that may act synergistically with L-arginine in enhancing exercise capacity.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 50-75 years, inclusive
* Ability to perform pulmonary function and exercise tests
* Willingness to take supplement powder for 3 weeks
* Ethical: Subject must sign the Institutional Review Board-approved written informed consent prior to he initiation of any study specific procedures or randomization. A subject will be excluded for any condition that might compromise the ability to give truly informed consent for participation in the study.

Exclusion Criteria:

* Existing pulmonary or cardiovascular disease
* Previous cardiac surgery
* Not able to tolerate breathing through mouthpiece for up to 20 minutes
* Musculoskeletal disease that would limit exercise

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-10; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Arginine and antioxidant supplements, as compared with placebo will improve exercise performance | 3 weeks

SECONDARY OUTCOMES:
Arginine and antioxidant Supplements improve maximal oxygen uptake and anaerobic threshold | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States